CLINICAL TRIAL: NCT00365963
Title: Clinician Integration Study
Brief Title: Web-based Intervention for Lung Cancer Patients and Their Informal Caregivers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2003-191X; 5P50CA095817-03 (NIH); CC04315 (Other: University of Wisconsin Carbone Cancer Center); 2003-191 (Other: Institutional Review Board); A195000 (Other: UW Madison); ENGR/INDUSTRIAL ENGR (Other: UW Madison)
Record Dates: First submitted 2006-08-16; First posted 2006-08-18 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2016-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: lung cancer, caregivers, support, resources, education
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

INTERVENTIONS:
Device: Comprehensive Health Enhancement Support System — computer based support and education

SUMMARY:
The purpose of this study is to find out if patients with lung cancer and their main informal caregiver (person providing physical, emotional, or financial support) are helped by getting information, support, and decision making tools through a computer system called CHESS(the Comprehensive Health Enhancement Support System)

DETAILED DESCRIPTION:
Many patients and their family/friends use the internet for obtaining information regarding the cancer diagnosis and treatment. In this study, the main caregiver of patients with advance (stage III or IV) non-small cell lung cancer is provided with a computer and internet access. Approximately one-half of the participants will also receive CHESS.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small Cell Lung Cancer (Stage III or Stage IV)
* Needs to have a "caregiver" - a spouse, partner, family member, or friend providing emotional, physical, and/or financial support - to participate with the patient.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Caregiver affect and adjustment | 1 year post patient death

SECONDARY OUTCOMES:
Clinician-Patient-Caregiver Communication | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — Center for Health Systems Research and Analysis
Locations (1):
- University of Wisconsin- Madison 610 Walnut St, WARF 1109A, Madison, Wisconsin, United States

REFERENCES:
- [Result] Gustafson DH, DuBenske LL, Atwood AK, Chih MY, Johnson RA, McTavish F, Quanbeck A, Brown RL, Cleary JF, Shah D. Reducing Symptom Distress in Patients With Advanced Cancer Using an e-Alert System for Caregivers: Pooled Analysis of Two Randomized Clinical Trials. J Med Internet Res. 2017 Nov 14;19(11):e354. doi: 10.2196/jmir.7466. PMID 29138131
- [Derived] DuBenske LL, Gustafson DH, Namkoong K, Hawkins RP, Atwood AK, Brown RL, Chih MY, McTavish F, Carmack CL, Buss MK, Govindan R, Cleary JF. CHESS improves cancer caregivers' burden and mood: results of an eHealth RCT. Health Psychol. 2014 Oct;33(10):1261-72. doi: 10.1037/a0034216. Epub 2013 Nov 18. PMID 24245838
- [Derived] Chih MY, DuBenske LL, Hawkins RP, Brown RL, Dinauer SK, Cleary JF, Gustafson DH. Communicating advanced cancer patients' symptoms via the Internet: a pooled analysis of two randomized trials examining caregiver preparedness, physical burden, and negative mood. Palliat Med. 2013 Jun;27(6):533-43. doi: 10.1177/0269216312457213. Epub 2012 Sep 17. PMID 22988042
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/